CLINICAL TRIAL: NCT01387815
Title: Canadian Humira Post Marketing Observational Epidemiological Study: Assessing Effectiveness in Psoriasis
Acronym: Complete-PS
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Cato Research (Industry); JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-678
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Psoriasis
Keywords: Effectiveness; Psoriasis; Observational; Prospective; Adalimumab; Traditional Systemic Agents; Topical Agents; Comparative
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Topical/Traditional Systemic Agent: Participants who initiated treatment with a new topical agent that was not used before or already being treated with topical agent and not responding, thereby requiring a change of treatment type, frequency, or dose and all participants who initiated treatment with a new systemic agent that was not used before alone or in combination with topical agents.
- Adalimumab: Participants treated with adalimumab alone or in combination with topical agents.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab administered by subcutaneous injection.
  Other Names: Humira
  Groups: Adalimumab

SUMMARY:
This was a Canadian post-marketing observational study (PMOS) utilizing a prospective cohort design that compared the real - life effectiveness of adalimumab to topical and traditional systemic agents in the management of psoriasis and its impact on the patient's quality of life and societal burden of illness.

DETAILED DESCRIPTION:
This was a Canadian post-marketing observational study (PMOS) utilizing a prospective cohort design. Participants were entered into one of two study cohorts (adalimumab cohort or topical/traditional systemic cohort) at the time of change of their psoriasis treatment for any reason and were followed for a maximum of 24 months with recommended assessments at 3, 6, 12, 18 and 24 months after baseline. Treatment of the participants and follow up were according to the physician's judgment, regional regulations, and the product monograph. Off-label use was not permitted, and these participants were not included in the study. Dose changes including escalation were allowed as per the physician's judgment for participants that were treated as per indication when they were enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Active moderate or severe plaque psoriasis according to the judgment of the treating physician.
* The treating physician has decided to change the current treatment or add additional treatments for any reason including but not limited to inadequate response, intolerance, sub-optimal compliance or participant preference.

Exclusion Criteria:

* Had currently participated in another prospective study with similar objectives.
* Participant could not or would not sign informed consent.
* Presence of other condition that, in the opinion of the treating physician, prohibits the participant from participating in the study or obscured the assessment of the treatment of plaque psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving treatment for psoriasis with adalimumab (alone or in combination with topical agents) or, either a topical (new, not used before or being treated and not responding) or, a traditional systemic agent (not used before alone or in combination with topical agents).
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2011-08-16 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (36):
- Canada (36):
  - Kirk Barber Research, CA /ID# 57722, Calgary, Alberta
  - Richmond Road Diagnostic Treat /ID# 70913, Calgary, Alberta
  - Institute for Skin Advancement /ID# 66782, Calgary, Alberta
  - Thomas Nakatsui P.C. /ID# 55080, Edmonton, Alberta
  - Alberta DermaSurgery Centre /ID# 75513, Edmonton, Alberta
  - Wellington Medical Clinic Ltd. /ID# 55083, Nanaimo, British Columbia
  - Percuro Clinical Research, Ltd /ID# 54563, Victoria, British Columbia
  - Jason Ronald Sneath Medical Co /ID# 138026, Brandon, Manitoba
  - Winnipeg Clinic, Manitoba, CA /ID# 56865, Winnipeg, Manitoba
  - Maritime Medical Reseach Cente /ID# 128775, Bathurst, New Brunswick
  - Dr. Irina Turchin PC Inc. /ID# 66029, Fredericton, New Brunswick
  - Dermatologue Inc. /ID# 76074, Moncton, New Brunswick
  - Douglas N. Keeling MD Dermatol /ID# 55098, Quispamsis, New Brunswick
  - Karma Clinical Trials /ID# 55101, St. John's, Newfoundland and Labrador
  - Nexus Clinical Research /ID# 56403, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Resea /ID# 46353, Halifax, Nova Scotia
  - SimcoDerm Medical and Surgical /ID# 96915, Barrie, Ontario
  - Kingsway Clinical Research /ID# 97255, Etobicoke, Ontario
  - Giroux, Sudbury, CA /ID# 55128, Greater Sudbury, Ontario
  - Dermatrials Research /ID# 124138, Hamilton, Ontario
  - Dr. Wei Jing Loo Medicine Prof /ID# 127546, London, Ontario
  - Lynderm Research Inc. /ID# 63206, Markham, Ontario
  - Toronto Regional Wound Healing /ID# 55135, Mississauga, Ontario
  - Dr. Anna Hinek Medicine Prof /ID# 148305, Mississauga, Ontario
  - Oakville Derma and Laser, CA /ID# 55130, Oakville, Ontario
  - Dr. Melinda Gooderham Medicine /ID# 54566, Peterborough, Ontario
  - York Dermatology Center /ID# 127786, Richmond Hill, Ontario
  - Specialized Dermatology Inc. /ID# 64031, St. Catharines, Ontario
  - Lori Shapiro Medicine Prof Inc /ID# 55126, Thornhill, Ontario
  - Toronto Dermatology Centre /ID# 55127, Toronto, Ontario
  - Dr. Isabelle Delorme Inc. /ID# 57791, Drummondville, Quebec
  - Dre. Angelique Gagne-Henley /ID# 125204, Montreal, Quebec
  - Dr. Loukia-Maria Mitsos /ID# 124156, Pierrefonds, Quebec
  - Dermatologie Sima Inc. /ID# 54922, Verdun, Quebec
  - Dr. Beatrice Wang /ID# 63242, Westmount, Quebec
  - Royal Univ. Hosp, Saskatoon,CA /ID# 74613, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 662 patients enrolled, the Safety Analysis Set included all who signed the inform consent and received at least 1 dose of study medication (N = 658) and the Intent-to-Treat Population included all who signed informed consent, met the inclusion / exclusion criteria, and received at least 1 dose of study medication (N = 595).
Period: Overall Study
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Started (Participant flow shows intent to treat (ITT) population (595) vs. enrolled (662).) | 302 | 293
Completed | 162 | 189
Not Completed | 140 | 104

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the intent to treat (ITT) population (595) vs. enrolled (662).
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab | Total
Number analyzed (Participants) | 302 | 293 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (15.06) | 48.2 (13.59) | 49.3 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 116 | 241
  Male | 177 | 177 | 354
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 262 | 255 | 517
  Black or African American | 1 | 3 | 4
  Asian | 23 | 26 | 49
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 4 | 0 | 4
  Other | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Physician Global Assessment (PGA) Score ≤1 at Month 6
Description: The Physician global assessment (PGA) score is an assessment by the investigator of the overall disease severity at the time of evaluation. The PGA uses a 6-point scale. The degree of overall lesion severity was evaluated using the following categories:
  * 0 (Clear): No evidence of scaling or plaque elevation; erythema may be present;
  * 1 (Minimal): scaling may be present, up to moderate erythema, minimal plaque elevation;
  * 2 (Mild): Fine scaling, up to moderate erythema, slight plaque elevation;
  * 3 (Moderate): Coarse scale dominates, moderate erythema, moderate plaque elevation;
  * 4 (Severe): Coarse non-tenacious scale dominates, severe erythema, marked plaque elevation;
  * 5 (Very Severe): Very coarse thick tenacious scale predominates, very severe erythema, severe plaque elevation.
  A higher score indicates greater disease severity. Percentages based on the total number of intent to treat (ITT) participants who attended each visit.
Time Frame: Month 6
Population: ITT population: all participants who signed informed consent, met inclusion/exclusion criteria, and received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants | 31.4 | 56.3
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Comparison does not include missing; Test type: Other; p < 0.001, Chi-squared

2. Secondary Outcome: Time to Achieving PGA ≤ 1
Description: The PGA is an assessment by the investigator of the overall disease severity at the time of evaluation. The PGA uses a 6-point scale. The degree of overall lesion severity was evaluated using the following categories:
  * 0 (Clear): No evidence of scaling or plaque elevation; erythema may be present;
  * 1 (Minimal): scaling may be present, up to moderate erythema, minimal plaque elevation;
  * 2 (Mild): Fine scaling, up to moderate erythema, slight plaque elevation;
  * 3 (Moderate): Coarse scale dominates, moderate erythema, moderate plaque elevation;
  * 4 (Severe): Coarse non-tenacious scale dominates, severe erythema, marked plaque elevation;
  * 5 (Very Severe): Very coarse thick tenacious scale predominates, very severe erythema, severe plaque elevation.
  A higher score indicates greater disease severity.
Time Frame: Baseline, Month 3, Month 6, Month 12, Month 18, and Month 24
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
Months | 13.3 [11.8 to 22.0] | 5.7 [4.4 to 6.0]
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p < 0.001, Log Rank

3. Secondary Outcome: PGA≤1: Percentage of Participants at Month 3
Description: The PGA is an assessment by the investigator of the overall disease severity at the time of evaluation. The PGA uses a 6-point scale. The degree of overall lesion severity was evaluated using the following categories:
  * 0 (Clear): No evidence of scaling or plaque elevation; erythema may be present;
  * 1 (Minimal): scaling may be present, up to moderate erythema, minimal plaque elevation;
  * 2 (Mild): Fine scaling, up to moderate erythema, slight plaque elevation;
  * 3 (Moderate): Coarse scale dominates, moderate erythema, moderate plaque elevation;
  * 4 (Severe): Coarse non-tenacious scale dominates, severe erythema, marked plaque elevation;
  * 5 (Very Severe): Very coarse thick tenacious scale predominates, very severe erythema, severe plaque elevation.
  A higher score indicates greater disease severity. Percentages based on the total number of ITT participants who attended each visit.
Time Frame: Month 3
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants | 19.0 | 47.5
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p < 0.001, Chi-squared

4. Secondary Outcome: PGA≤1: Percentage of Participants at Month 12
Description: as for outcome 3
Time Frame: Month 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants | 34.5 | 57.3
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p < 0.001, Chi-squared

5. Secondary Outcome: PGA≤1: Percentage of Participants at Month 18
Description: as for outcome 3
Time Frame: Month 18
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants | 35.7 | 61.3
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p < 0.001, Chi-squared

6. Secondary Outcome: PGA≤1: Percentage of Participants at Month 24
Description: as for outcome 3
Time Frame: Month 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants | 37.5 | 56.7
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p < 0.001, Chi-squared

7. Secondary Outcome: Psoriasis and Arthritis Screening Questionnaire (PASQ) Total Score: Change From Baseline to Month 3
Description: PASQ is an 11-item tool that ascertains self-reported presence of joint pain and swelling by the participant. The PASQ questionnaire consists of 10 questions for which a positive and negative response are assigned a score of 1 or 2, and 0, respectively. The maximum score is 10. In addition, participants were also asked to indicate on a diagram where they experienced joint swelling or pain. The diagram was scored 0, 1, 3, or 5, depending on the distribution of the participants' markings. The final composite score for the PASQ ranges from 0 to a maximum of 15. A decrease indicates improvement.
Time Frame: Baseline, Month 3
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 189 | 184
score on a scale | 6.3 (4.28) | 7.6 (4.48)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.003, t-test, 2 sided

8. Secondary Outcome: PASQ Total Score: Change From Baseline to Month 6
Description: as for outcome 7
Time Frame: Baseline, Month 6
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 161 | 172
score on a scale | 6.3 (4.35) | 7.5 (4.48)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.016, t-test, 2 sided

9. Secondary Outcome: PASQ Total Score: Change From Baseline to Month 12
Description: as for outcome 7
Time Frame: Baseline, Month 12
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 139 | 147
score on a scale | 6.6 (4.46) | 7.6 (4.25)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.060, t-test, 2 sided

10. Secondary Outcome: PASQ Total Score: Change From Baseline to Month 18
Description: as for outcome 7
Time Frame: Baseline, Month 18
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 113 | 114
score on a scale | 6.9 (4.05) | 7.9 (4.22)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.056, t-test, 2 sided

11. Secondary Outcome: PASQ Total Score: Change From Baseline to Month 24
Description: as for outcome 7
Time Frame: Baseline, Month 24
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 108 | 111
score on a scale | 7.2 (4.49) | 7.4 (4.21)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.755, t-test, 2 sided

12. Secondary Outcome: Body Surface Area of Psoriasis Involvement: Change From Baseline to Month 6
Description: The Body Surface Area (BSA) is an indicator of disease severity and the affected area is expressed as a percentage of the total body surface area.The BSA affected by psoriasis was measured by the physician selecting the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus 5 digits was to be assumed to be approximately equivalent to 1% BSA. Measurement of the total area of involvement by the physician was aided by imagining if scattered plaques were moved so that they were next to each other and then estimated the total area involved. A decrease in BSA affected by psoriasis indicates improvement.
Time Frame: Baseline, Month 6
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: percentage estimated body surface area
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 195 | 211
percentage estimated body surface area | 6.4 (7.30) | 4.9 (10.14)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.091, t-test, 2 sided

13. Secondary Outcome: BSA of Psoriasis Involvement: Change From Baseline to Month 12
Description: The BSA is an indicator of disease severity and the affected area is expressed as a percentage of the total body surface area.The BSA affected by psoriasis was measured by the physician selecting the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus 5 digits was to be assumed to be approximately equivalent to 1% BSA. Measurement of the total area of involvement by the physician was aided by imagining if scattered plaques were moved so that they were next to each other and then estimated the total area involved. A decrease in BSA affected by psoriasis indicates improvement.
Time Frame: Baseline, Month 12
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: percentage estimated body surface area
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 177 | 195
percentage estimated body surface area | 5.4 (7.29) | 4.1 (8.25)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.106, t-test, 2 sided

14. Secondary Outcome: BSA of Psoriasis Involvement: Change From Baseline to Month 18
Description: as for outcome 13
Time Frame: Baseline, Month 18
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: percentage estimated body surface area
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 149 | 167
percentage estimated body surface area | 5.1 (6.03) | 3.1 (5.58)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.003, t-test, 2 sided

15. Secondary Outcome: BSA of Psoriasis Involvement: Change From Baseline to Month 24
Description: as for outcome 13
Time Frame: Baseline, Month 24
Population: ITT population of participants who were available for assessment at this visit.
Measure: Mean (Standard Deviation); unit: percentage estimated body surface area
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 143 | 166
percentage estimated body surface area | 6.3 (10.37) | 3.7 (6.63)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.008, t-test, 2 sided

16. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity Based on a Visual Analog Scale (VAS): Change From Baseline to Month 3
Description: Patient Global Assessment of disease activity (PtGA) was assessed using a visual analog scale (VAS) where 0 indicates doing very well with respect to arthritis and/or skin psoriasis and a value of 100 indicates doing very poorly.
Time Frame: Baseline, Month 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 215
units on a scale | 37.3 (27.13) | 32.8 (27.72)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.083, t-test, 2 sided

17. Secondary Outcome: PtGA of Disease Activity Based on a VAS: Change From Baseline to Month 6
Description: PtGA of disease activity was assessed using a VAS where 0 indicates doing very well with respect to arthritis and/or skin psoriasis and a value of 100 indicates doing very poorly.
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 188 | 201
units on a scale | 31.8 (27.44) | 29.9 (28.28)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.495, t-test, 2 sided

18. Secondary Outcome: PtGA of Disease Activity Based on a VAS: Change From Baseline to Month 12
Description: as for outcome 17
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 179 | 180
units on a scale | 32.9 (27.33) | 28.2 (27.07)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.097, t-test, 2 sided

19. Secondary Outcome: PtGA of Disease Activity Based on a VAS: Change From Baseline to Month 18
Description: as for outcome 17
Time Frame: Baseline, Month 18
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 144 | 153
units on a scale | 30.2 (27.61) | 21.8 (24.89)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.006, t-test, 2 sided

20. Secondary Outcome: PtGA of Disease Activity Based on a VAS: Change From Baseline to Month 24
Description: as for outcome 17
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 141 | 143
units on a scale | 31.9 (27.60) | 25.1 (26.65)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.037, t-test, 2 sided

21. Secondary Outcome: Dermatology Quality of Life Index (DLQI) Total Score: Change From Baseline to Month 3
Description: The Dermatology Quality of Life Index (DLQI) is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 1 to 30, where 0-1 = no effect on participant's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on participant's life. The higher the score, the more the participant's quality of life is impaired. A 5-point change from baseline is considered a clinically important difference.
Time Frame: Baseline, Month 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 219 | 215
score on a scale | 6.5 (6.31) | 5.4 (6.18)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.084, t-test, 2 sided

22. Secondary Outcome: DLQI Total Score: Change From Baseline to Month 6
Description: The DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 1 to 30, where 0-1 = no effect on participant's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on participant's life. The higher the score, the more the participant's quality of life is impaired. A 5-point change from baseline is considered a clinically important difference.
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 185 | 197
score on a scale | 5.3 (6.01) | 4.3 (6.00)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.090, t-test, 2 sided

23. Secondary Outcome: DLQI Total Score: Change From Baseline to Month 12
Description: as for outcome 22
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 174 | 179
score on a scale | 5.1 (5.73) | 3.9 (5.66)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.059, t-test, 2 sided

24. Secondary Outcome: DLQI Total Score: Change From Baseline to Month 18
Description: as for outcome 22
Time Frame: Baseline, Month 18
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 141 | 149
score on a scale | 4.0 (5.05) | 2.5 (3.70)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.004, t-test, 2 sided

25. Secondary Outcome: DLQI Total Score: Change From Baseline to Month 24
Description: as for outcome 22
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 143 | 141
score on a scale | 4.3 (5.15) | 3.3 (5.03)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.115, t-test, 2 sided

26. Secondary Outcome: Time to Achieving DLQI ≤1
Description: as for outcome 22
Time Frame: Baseline, Month 3, Month 6, Month 12, Month 18, and Month 24
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 277 | 267
Months | 17.7 [11.5 to NA] — Upper limit could not be calculated. | 8.2 [6.3 to 12.0]
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.002, Log Rank

27. Secondary Outcome: DLQI ≤1: Percentage of Participants at Month 3
Description: The DLQI is a 10-question questionnaire that asks the participant to evaluate the degree that psoriasis has affected their quality of life in the last week and includes 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). Responses to each domain are not relevant (0), not at all (0), a little (1), a lot (2), and very much (3). The DLQI is calculated by summing the scores of the questions and ranges from 1 to 30, where 0-1 = no effect on participant's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on participant's life. The higher the score, the more the participant's quality of life is impaired. A 5-point change from baseline is considered a clinically important difference. Percentage based on the total number of ITT participants who attended each visit.
Time Frame: Month 3
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants
  No effect at all on patient's life (0-1) | 18.2 | 31.1
  Small effect on patient's life (2-5) | 33.2 | 21.4
  Moderate effect on patient's life (6-10) | 19.0 | 15.6
  Very large effect on patient's life (21-30) | 13.4 | 12.8
  Extremely large effect on patient's life (21-30) | 4.9 | 2.7
  Missing | 11.3 | 16.3
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Comparison does not include the "Missing" category; Test type: Other; p = 0.002, Chi-squared

28. Secondary Outcome: DLQI ≤1: Percentage of Participants at Month 6
Description: as for outcome 27
Time Frame: Month 6
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants
  No effect at all on patient's life (0-1) | 26.5 | 39.3
  Small effect on patient's life (2-5) | 28.7 | 19.8
  Moderate effect on patient's life (6-10) | 13.5 | 10.1
  Very large effect on patient's life (21-30) | 11.2 | 8.5
  Extremely large effect on patient's life (21-30) | 3.1 | 2.0
  Missing | 17.0 | 20.2
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other — Comparison does not include the "Missing" category; p = 0.017, Chi-squared

29. Secondary Outcome: DLQI ≤1: Percentage of Participants at Month 12
Description: as for outcome 27
Time Frame: Month 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants
  No effect at all on patient's life (0-1) | 28.2 | 37.9
  Small effect on patient's life (2-5) | 27.2 | 24.2
  Moderate effect on patient's life (6-10) | 15.0 | 7.5
  Very large effect on patient's life (21-30) | 12.1 | 6.2
  Extremely large effect on patient's life (21-30) | 1.9 | 3.1
  Missing | 15.5 | 21.1
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.010, Chi-squared — Comparison does not include the "Missing" category

30. Secondary Outcome: DLQI ≤1: Percentage of Participants at Month 18
Description: as for outcome 27
Time Frame: Month 18
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants
  No effect at all on patient's life (0-1) | 35.7 | 45.7
  Small effect on patient's life (2-5) | 25.7 | 15.6
  Moderate effect on patient's life (6-10) | 12.9 | 11.1
  Very large effect on patient's life (21-30) | 7.0 | 2.0
  Extremely large effect on patient's life (21-30) | 1.2 | 0.5
  Missing | 17.5 | 25.1
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Comparison does not include the "Missing" category; Test type: Other; p = 0.015, Chi-squared

31. Secondary Outcome: DLQI ≤1: Percentage of Participants at Month 24
Description: as for outcome 27
Time Frame: Month 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 302 | 293
percentage of participants
  No effect at all on patient's life (0-1) | 34.5 | 38.1
  Small effect on patient's life (2-5) | 27.4 | 20.1
  Moderate effect on patient's life (6-10) | 12.5 | 9.8
  Very large effect on patient's life (21-30) | 9.5 | 2.6
  Extremely large effect on patient's life (21-30) | 1.2 | 2.1
  Missing | 14.9 | 27.3
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Comparison does not include the "Missing" category; Test type: Other; p = 0.060, Chi-squared

32. Secondary Outcome: Beck Depression Inventory II (BDI-II): Change From Baseline to Month 6
Description: The Beck Depression inventory assesses the presence and severity of depression and responsiveness to treatment. It consists of 21 items converging on 2 scales measuring somatic and affective components of depression. The questions assess hopelessness and irritability, cognition such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and loss of interest in sex.
  The total score ranges from a minimum of 0 to a maximum of 63 with the following suggested score interpretations: minimal range = 0-13, mild depression = 14-19, moderate depression = 20-28, and severe depression = 29-63.
  The higher the score, the greater the severity of the depression.
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 184 | 195
score on a scale | 7.8 (8.95) | 7.2 (7.80)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.501, t-test, 2 sided

33. Secondary Outcome: BDI-II: Change From Baseline to Month 12
Description: as for outcome 32
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 177 | 178
score on a scale | 7.5 (8.06) | 7.3 (7.72)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.807, t-test, 2 sided

34. Secondary Outcome: BDI-II: Change From Baseline to Month 24
Description: as for outcome 32
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 140 | 142
score on a scale | 7.2 (7.59) | 6.6 (7.51)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.479, t-test, 2 sided

35. Secondary Outcome: Medical Outcomes Study Short Form-12 Health Status Survey (SF-12) Mental Component Summary (MCS) Score: Change From Baseline to Month 6
Description: The Medical Outcomes Study Short Form 12 (SF-12) questionnaire is a shortened form (12 items) of the SF-36 Health Survey generic quality of life questionnaire that assesses eight health concepts: 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality (energy and fatigue); 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health (psychological distress and well-being). Items 5-8 comprise the mental component of the SF-12. Scores on each item were summed and averaged (MCS Score; range = 0-100); a positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 119 | 120
score on a scale | 49.8 (10.43) | 49.7 (10.08)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.918, t-test, 2 sided

36. Secondary Outcome: SF-12 MCS Score: Change From Baseline to Month 12
Description: The SF-12 questionnaire is a shortened form (12 items) of the SF-36 Health Survey generic quality of life questionnaire that assesses eight health concepts: 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality (energy and fatigue); 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health (psychological distress and well-being). Items 5-8 comprise the mental component of the SF-12. Scores on each item were summed and averaged (MCS Score; range = 0-100); a positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 123 | 113
score on a scale | 48.9 (11.37) | 49.6 (9.99)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.609, t-test, 2 sided

37. Secondary Outcome: SF-12 MCS Score: Change From Baseline to Month 24
Description: as for outcome 36
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 121 | 114
score on a scale | 50.2 (10.92) | 51.3 (8.93)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.367, t-test, 2 sided

38. Secondary Outcome: SF-12 Physical Component Summary (PCS) Score: Change From Baseline to Month 6
Description: The SF-12 questionnaire is a shortened form (12 items) of the SF-36 Health Survey generic quality of life questionnaire that assesses eight health concepts: 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality (energy and fatigue); 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health (psychological distress and well-being). Items 1-4 comprise the physical component of the SF-12. Scores on each item were summed and averaged (PCS Score; range = 0-100); a positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 119 | 120
score on a scale | 48.2 (10.14) | 47.3 (10.35)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.521, t-test, 2 sided

39. Secondary Outcome: SF-12 PCS Score: Change From Baseline to Month 12
Description: as for outcome 38
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 123 | 113
score on a scale | 47.3 (10.93) | 47.0 (10.40)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.793, t-test, 2 sided

40. Secondary Outcome: SF-12 PCS Score: Change From Baseline to Month 24
Description: as for outcome 38
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 121 | 114
score on a scale | 47.8 (9.81) | 48.8 (9.81)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.442, t-test, 2 sided

41. Secondary Outcome: Work Limitation Questionnaire (WLQ) Total Score: Change From Baseline to Month 6
Description: The Work Limitation Questionnaire (WLQ) is a self-administered questionnaire comprised of 25 questions.
  The WLQ evaluates the participant's overall ability to work in the last two weeks. It comprises 25 questions each with a range of 100% ('all of the time') to 0% ('none of the time') where 6 represents non-applicability to the patient's line of work.
  The WLQ Productivity Loss Score indicates the percentage decrement in work output due to health problems. The WLQ Productivity Loss score is based on a weighted sum of the scores from the 4 WLQ scales (Time, Physical, Mental-Interpersonal, and Output). The resulting score (known as the WLQ Index) is in the form of the natural log of work productivity. The final step needed to generate the WLQ Productivity Loss Score is to convert the WLQ Index score to a percentage. The higher the score, the greater the work limitation.
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 117 | 138
score on a scale | 12.4 (15.67) | 14.0 (16.44)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.434, t-test, 2 sided

42. Secondary Outcome: WLQ Total Score: Change From Baseline to Month 12
Description: The WLQ is a self-administered questionnaire comprised of 25 questions. The WLQ evaluates the participant's overall ability to work in the last two weeks. It comprises 25 questions each with a range of 100% ('all of the time') to 0% ('none of the time') where 6 represents non-applicability to the patient's line of work.
  The WLQ Productivity Loss Score indicates the percentage decrement in work output due to health problems. The WLQ Productivity Loss score is based on a weighted sum of the scores from the 4 WLQ scales (Time, Physical, Mental-Interpersonal, and Output). The resulting score (known as the WLQ Index) is in the form of the natural log of work productivity. The final step needed to generate the WLQ Productivity Loss Score is to convert the WLQ Index score to a percentage. The higher the score, the greater the work limitation.
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 107 | 109
score on a scale | 13.5 (15.45) | 14.2 (17.52)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.752, t-test, 2 sided

43. Secondary Outcome: WLQ Total Score: Change From Baseline to Month 24
Description: as for outcome 42
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 84 | 91
score on a scale | 12.1 (15.51) | 10.4 (15.86)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.469, t-test, 2 sided

44. Secondary Outcome: WLQ Productivity Loss Score: Change From Baseline to Month 6
Description: as for outcome 42
Time Frame: Baseline, Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 117 | 138
score on a scale | 3.2 (4.19) | 3.6 (4.25)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.419, t-test, 2 sided

45. Secondary Outcome: WLQ Productivity Loss Score: Change From Baseline to Month 12
Description: as for outcome 42
Time Frame: Baseline, Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 107 | 109
score on a scale | 3.5 (4.07) | 3.7 (4.73)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.695, t-test, 2 sided

46. Secondary Outcome: WLQ Productivity Loss Score: Change From Baseline to Month 24
Description: as for outcome 42
Time Frame: Baseline, Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 84 | 91
score on a scale | 3.1 (4.16) | 2.7 (4.11)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.452, t-test, 2 sided

47. Secondary Outcome: Healthcare Resource Utilization (HCRU): Number of Participants With Insurance for Prescription Medication at Month 6
Description: Participants were asked at Month 6, Month 12, and Month 24 about having insurance for prescription medication (and type of insurance) and their utilization of healthcare resources within the 4 weeks prior to study visits: seeking health care for AS, including extra/unscheduled office visits to their study doctor (and number of visits among those reporting ≥1 visit), visits to another doctor (and number of visits among those reporting ≥1 visit), visits to healthcare professional (and number of visits among those reporting ≥1 visit), visits to hospital emergency room (and number of visits among those reporting ≥1 visit), use of ambulant service, complementary/alternate therapy visits (and number of visits among those reporting ≥1 visit), hospital admissions (and length of hospital stay), ICU admissions, over the counter medications, payments for healthcare professionals, medical procedures or laboratory tests, medical devices, health care or extra help at home, and transportation costs.
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants | 156 | 177
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.008, t-test, 2 sided

48. Secondary Outcome: HCRU: Number of Participants With Insurance for Prescription Medication at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants | 148 | 157
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.181, t-test, 2 sided

49. Secondary Outcome: HCRU: Number of Participants With Insurance for Prescription Medication at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants | 112 | 121
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.252, t-test, 2 sided

50. Secondary Outcome: HCRU: Number of Participants by Type of Insurance for Prescription Medication at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population of participants who were available for assessment at this visit and answered "yes" to question of having insurance for prescription medication. Note: One patient may have had more than one medical insurance; therefore, the total of the rows will not match the number analyzed.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 156 | 177
participants
  RAMQ | 14 | 8
  Federal Government | 8 | 12
  OHIP | 17 | 29
  Blue Cross | 26 | 28
  Other | 74 | 74
  Missing: Insurer name not provided | 30 | 42

51. Secondary Outcome: HCRU: Number of Participants by Type of Insurance for Prescription Medication at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: as for outcome 50
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 148 | 157
participants
  RAMQ | 13 | 6
  Federal Government | 6 | 6
  CSST | 1 | 0
  OHIP | 26 | 24
  Blue Cross | 23 | 29
  Other | 66 | 76
  Missing: Insurer name not provided | 27 | 38

52. Secondary Outcome: HCRU: Number of Participants by Type of Insurance for Prescription Medication at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: as for outcome 50
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 112 | 121
participants
  RAMQ | 8 | 5
  Federal Government | 7 | 6
  OHIP | 16 | 27
  Blue Cross | 18 | 24
  Other | 51 | 48
  Missing: Insurer name not provided | 24 | 24

53. Secondary Outcome: HCRU: Number of Participants Seeking Health Care in the Past 4 Weeks for Ankylosing Spondylitis (AS) at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 95 | 86
  No | 82 | 101
  Missing | 46 | 60
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.143, Chi-squared

54. Secondary Outcome: HCRU: Number of Participants Seeking Health Care in the Past 4 Weeks for AS at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 89 | 81
  No | 81 | 88
  Missing | 36 | 58
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.415, Chi-squared

55. Secondary Outcome: HCRU: Number of Participants Seeking Health Care in the Past 4 Weeks for AS at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 57 | 55
  No | 71 | 78
  Missing | 40 | 61
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.604, Chi-squared

56. Secondary Outcome: HCRU: Number of Participants Making Extra or Unscheduled Visits the (Office/Clinic) of the Study Doctor for AS at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 7 | 5
  No | 71 | 76
  Missing | 145 | 166
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.504, Fisher Exact

57. Secondary Outcome: HCRU: Number of Participants Making Extra or Unscheduled Visits the (Office/Clinic) of the Study Doctor for AS at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 7 | 7
  No | 73 | 69
  Missing | 126 | 151
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.920, Chi-squared

58. Secondary Outcome: HCRU: Number of Participants Making Extra or Unscheduled Visits the (Office/Clinic) of the Study Doctor for AS at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 3 | 2
  No | 51 | 49
  Missing | 114 | 143
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p > 0.999, Fisher Exact

59. Secondary Outcome: HCRU: Number of Extra or Unscheduled Visits the (Office/Clinic) of the Study Doctor for AS at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 7 | 3
office visits | 1.9 (1.46) | 1.3 (0.58)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.575, Chi-squared

60. Secondary Outcome: HCRU: Number of Extra or Unscheduled Visits the (Office/Clinic) of the Study Doctor for AS at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 3 | 1
office visits | 1.0 (0.00) | NA (NA) — There was only one participant to analyze, so a mean could not be calculated.

61. Secondary Outcome: HCRU: Number of Extra or Unscheduled Visits the (Office/Clinic) of the Study Doctor for AS at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 3 | 1
office visits | 7.0 (1.73) | NA (NA) — The mean could not be calculated because there was only one participant.

62. Secondary Outcome: HCRU: Number of Participants Making Visits to Another Physician at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 21 | 20
  No | 59 | 60
  Missing | 143 | 167
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.856, Chi-squared

63. Secondary Outcome: HCRU: Number of Participants Making Visits to Another Physician at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 18 | 14
  No | 58 | 55
  Missing | 130 | 158
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.623, Chi-squared

64. Secondary Outcome: HCRU: Number of Participants Making Visits to Another Physician at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 15 | 16
  No | 38 | 35
  Missing | 115 | 143
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.732, Chi-squared

65. Secondary Outcome: HCRU: Number of Visits to Another Physician at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 11 | 7
office visits | 1.4 (1.21) | 1.4 (0.53)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.896, t-test, 2 sided

66. Secondary Outcome: HCRU: Number of Visits to Another Physician at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 4 | 5
office visits | 2.0 (1.41) | 2.2 (2.17)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.879, t-test, 2 sided

67. Secondary Outcome: HCRU: Number of Visits to Another Physician at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 5 | 7
office visits | 1.2 (0.45) | 1.3 (0.49)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.763, t-test, 2 sided

68. Secondary Outcome: HCRU: Number of Participants Making Visits to a Healthcare Professional at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 15 | 12
  No | 61 | 59
  Missing | 147 | 176
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.657, Chi-squared

69. Secondary Outcome: HCRU: Number of Participants Making Visits to a Healthcare Professional at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 13 | 12
  No | 60 | 55
  Missing | 133 | 160
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.987, Chi-squared

70. Secondary Outcome: HCRU: Number of Participants Making Visits to a Healthcare Professional at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 2 | 10
  No | 49 | 39
  Missing | 117 | 145
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.011, Fisher Exact

71. Secondary Outcome: HCRU: Number of Visits to A Healthcare Professional at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 8 | 2
office visits | 1.3 (0.71) | 1.0 (0.00)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.351, t-test, 2 sided

72. Secondary Outcome: HCRU: Number of Visits to A Healthcare Professional at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 5 | 2
office visits | 1.8 (1.79) | 1.5 (0.71)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.835, t-test, 2 sided

73. Secondary Outcome: HCRU: Number of Visits to A Healthcare Professional at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: office visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 1 | 3
office visits | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed. | 1.3 (0.58)

74. Secondary Outcome: HCRU: Number of Participants Making Visits to a Hospital Emergency Room at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 3 | 4
  No | 83 | 77
  Missing | 137 | 166
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.714, Fisher Exact

75. Secondary Outcome: HCRU: Number of Participants Making Visits to a Hospital Emergency Room at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 4 | 5
  No | 82 | 73
  Missing | 120 | 149
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.737, Fisher Exact

76. Secondary Outcome: HCRU: Number of Participants Making Visits to a Hospital Emergency Room at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 2 | 3
  No | 52 | 51
  Missing | 114 | 140
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p > 0.999, Fisher Exact

77. Secondary Outcome: HCRU: Number of Visits to a Hospital Emergency Room at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 0 | 1
visits |  | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.

78. Secondary Outcome: HCRU: Number of Visits to a Hospital Emergency Room at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 1 | 1
visits | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed. | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.

79. Secondary Outcome: HCRU: Number of Visits to a Hospital Emergency Room at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 0 | 1
visits |  | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.

80. Secondary Outcome: HCRU: Number of Participants Making Use of an Ambulance Service at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 1 | 0
  No | 84 | 81
  Missing | 138 | 166
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p > 0.999, Fisher Exact

81. Secondary Outcome: HCRU: Number of Participants Making Use of an Ambulance Service at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 1 | 1
  No | 85 | 77
  Missing | 120 | 149
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p > 0.999, Fisher Exact

82. Secondary Outcome: HCRU: Number of Participants Making Use of an Ambulance Service at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  No | 54 | 54
  Missing | 114 | 140

83. Secondary Outcome: HCRU: Number of Participants Making Complementary/Alternate Therapy Visits at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 3 | 4
  No | 84 | 78
  Missing | 136 | 165
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.714, Fisher Exact

84. Secondary Outcome: HCRU: Number of Participants Making Complementary/Alternate Therapy Visits at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 6 | 4
  No | 76 | 73
  Missing | 124 | 150
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.747, Fisher Exact

85. Secondary Outcome: HCRU: Number of Participants Making Complementary/Alternate Therapy Visits at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 0 | 1
  No | 54 | 52
  Missing | 114 | 141
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.495, Fisher Exact

86. Secondary Outcome: HCRU: Number of Complementary/Alternate Therapy Visits at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 2 | 0
visits | 3.0 (1.41) |

87. Secondary Outcome: HCRU: Number of Complementary/Alternate Therapy Visits at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 1 | 1
visits | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed. | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.

88. Secondary Outcome: HCRU: Number of Complementary/Alternate Therapy Visits at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 0 | 0

89. Secondary Outcome: HCRU: Number of Participants Hospitalized in the Past 4 Weeks at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 3 | 1
  No | 177 | 186
  Missing | 43 | 60
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.364, Fisher Exact

90. Secondary Outcome: HCRU: Number of Participants Hospitalized in the Past 4 Weeks at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 3 | 3
  No | 167 | 172
  Missing | 36 | 52
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p > 0.999, Fisher Exact

91. Secondary Outcome: HCRU: Number of Participants Hospitalized in the Past 4 Weeks at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 3 | 5
  No | 130 | 132
  Missing | 35 | 57
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.723, Fisher Exact

92. Secondary Outcome: HCRU: Length of Hospital Stay for Those Participants Hospitalized at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 3 | 1
days | 8.3 (7.51) | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.

93. Secondary Outcome: HCRU: Length of Hospital Stay for Those Participants Hospitalized at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 1 | 3
days | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed. | 2.0 (1.00)

94. Secondary Outcome: HCRU: Length of Hospital Stay for Those Participants Hospitalized at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 1 | 1
days | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed. | 1 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.

95. Secondary Outcome: HCRU: Number of Participants Admitted to the Intensive Care Unit (ICU) in the Past 4 Weeks at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 1 | 0
  Missing | 222 | 247

96. Secondary Outcome: HCRU: Number of Participants Admitted to the ICU in the Past 4 Weeks at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 0 | 1
  Missing | 206 | 226

97. Secondary Outcome: HCRU: Number of Participants Admitted to the ICU in the Past 4 Weeks at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population. Data not collected.
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 0 | 0

98. Secondary Outcome: HCRU: Cost of Payment for Over the Counter Medications at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 86 | 86
dollars | 35.0 (77.82) | 8.7 (37.85)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.006, t-test, 2 sided

99. Secondary Outcome: HCRU: Cost of Payment for Over the Counter Medications at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 66 | 82
dollars | 17.8 (48.28) | 22.1 (73.15)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.672, t-test, 2 sided

100. Secondary Outcome: HCRU: Cost of Payment for Over the Counter Medications at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 49 | 63
dollars | 10.8 (21.43) | 17.3 (69.10)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.482, t-test, 2 sided

101. Secondary Outcome: HCRU: Cost of Payments to Healthcare Professionals at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 68 | 81
dollars | 4.0 (28.34) | 4.4 (25.12)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.938, t-test, 2 sided

102. Secondary Outcome: HCRU: Cost of Payments to Healthcare Professionals at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 63 | 77
dollars | 31.2 (147.48) | 3.5 (21.48)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.144, t-test, 2 sided

103. Secondary Outcome: HCRU: Cost of Payments to Healthcare Professionals at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 40 | 53
dollars | 7.9 (42.44) | 1.5 (10.99)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.360, t-test, 2 sided

104. Secondary Outcome: HCRU: Cost of Payments for Medical Procedures or Laboratory Tests at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 68 | 81
dollars | 2.0 (12.20) | 2.6 (19.35)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.808, t-test, 2 sided

105. Secondary Outcome: HCRU: Cost of Payments for Medical Procedures or Laboratory Tests at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 59 | 76
dollars | 0.0 (0.00) | 0.5 (3.61)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.208, t-test, 2 sided

106. Secondary Outcome: HCRU: Cost of Payments for Medical Procedures or Laboratory Tests at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 40 | 54
dollars | 0.4 (2.37) | 8.2 (42.50)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.184, t-test, 2 sided

107. Secondary Outcome: HCRU: Cost of Payments for Medical Devices at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 68 | 80
dollars | 0.00 (0.00) | 0.4 (3.35)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.305, t-test, 2 sided

108. Secondary Outcome: HCRU: Cost of Payments for Medical Devices at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 59 | 76
dollars | 0.0 (0.00) | 0.0 (0.00)

109. Secondary Outcome: HCRU: Cost of Payments for Medical Devices at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 41 | 54
dollars | 1.0 (4.36) | 1.5 (10.89)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.757, t-test, 2 sided

110. Secondary Outcome: HCRU: Cost of Payments for Health Care or Extra Help at Home at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 68 | 79
dollars | 5.9 (48.51) | 0.0 (0.00)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.321, t-test, 2 sided

111. Secondary Outcome: HCRU: Cost of Payments for Health Care or Extra Help at Home at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 59 | 77
dollars | 0.0 (0.00) | 1.4 (8.87)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.181, t-test, 2 sided

112. Secondary Outcome: HCRU: Cost of Payments for Health Care or Extra Help at Home at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 40 | 54
dollars | 2.5 (15.81) | 18.5 (136.08)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.395, t-test, 2 sided

113. Secondary Outcome: HCRU: Cost of Payments for Transportation at Month 6
Description: as for outcome 47
Time Frame: Month 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 84 | 92
dollars | 20.4 (59.74) | 14.7 (45.31)

114. Secondary Outcome: HCRU: Cost of Payments for Transportation at Month 12
Description: as for outcome 47
Time Frame: Month 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 74 | 87
dollars | 13.1 (31.69) | 15.5 (56.74)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.739, t-test, 2 sided

115. Secondary Outcome: HCRU: Cost of Payments for Transportation at Month 24
Description: as for outcome 47
Time Frame: Month 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 59 | 60
dollars | 22.1 (50.70) | 12.9 (44.53)
Statistical Analysis 1: Comparison: Topical/Traditional Systemic Agent vs Adalimumab; Test type: Other; p = 0.291, t-test, 2 sided

116. Secondary Outcome: Topical Treatment Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 3
Description: Psoriasis treatment compliance by the participant was assessed by a self-administered questionnaire and interview by the treating physician at Month 3, 6, 12, 18, and 24. Participants were asked to complete the baseline set of questionnaires while at the physician's office. Thereafter, participants completed the questionnaires themselves and either mailed them to the data management center or returned them to the treating physician. The questions included the number missed since the last visit of: applications for topical medication; phototherapy sessions; doses of traditional systemic agents; and adalimumab injections.
Time Frame: Month 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 126 | 53
doses | 2.8 (8.94) | 2.2 (11.66)

117. Secondary Outcome: Topical Treatment Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 6
Description: as for outcome 116
Time Frame: Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 107 | 58
doses | 4.8 (16.90) | 3.3 (16.58)

118. Secondary Outcome: Topical Treatment Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 12
Description: as for outcome 116
Time Frame: Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 91 | 50
doses | 3.8 (13.40) | 0.6 (4.24)

119. Secondary Outcome: Topical Treatment Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 18
Description: as for outcome 116
Time Frame: Month 18
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 59 | 57
doses | 5.0 (28.31) | 0.3 (1.99)

120. Secondary Outcome: Topical Treatment Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 24
Description: as for outcome 116
Time Frame: Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 62 | 50
doses | 0.2 (0.95) | 0.1 (0.71)

121. Secondary Outcome: Phototherapy Session Patient Reported Treatment Compliance: Number of Missed Sessions Since Last Visit Assessed at Month 3
Description: Phototherapy sessions for psoriasis compliance by the participant was assessed by a self administered questionnaire and interview by the treating physician at Month 3, 6, 12, 18, and 24 as part of the psoriasis treatment compliance questionnaire. Participants were asked to complete the baseline set of questionnaires while at the physician's office. Thereafter, participants completed the questionnaires themselves and either mailed them to the data management center or returned them to the treating physician.
Time Frame: Month 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 31 | 4
sessions | 3.3 (9.11) | 2.5 (3.79)

122. Secondary Outcome: Phototherapy Session Patient Reported Treatment Compliance: Number of Missed Sessions Since Last Visit Assessed at Month 6
Description: as for outcome 121
Time Frame: Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 20 | 3
sessions | 1.8 (4.18) | 4.7 (4.16)

123. Secondary Outcome: Phototherapy Session Patient Reported Treatment Compliance: Number of Missed Sessions Since Last Visit Assessed at Month 12
Description: as for outcome 121
Time Frame: Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 22 | 3
sessions | 1.6 (3.24) | 1.3 (2.31)

124. Secondary Outcome: Phototherapy Session Patient Reported Treatment Compliance: Number of Missed Sessions Since Last Visit Assessed at Month 18
Description: as for outcome 121
Time Frame: Month 18
Population: ITT population
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 15 | 3
sessions | 0.3 (1.05) | 2.7 (3.06)

125. Secondary Outcome: Phototherapy Session Patient Reported Treatment Compliance: Number of Missed Sessions Since Last Visit Assessed at Month 24
Description: as for outcome 121
Time Frame: Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 15 | 2
sessions | 1.1 (2.40) | 10.0 (0.00)

126. Secondary Outcome: Traditional Systemic Agent Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 3
Description: as for outcome 116
Time Frame: Month 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 135 | 22
doses | 2.7 (10.10) | 0.0 (0.21)

127. Secondary Outcome: Traditional Systemic Agent Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 6
Description: as for outcome 116
Time Frame: Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 107 | 18
doses | 3.0 (12.98) | 0.1 (0.47)

128. Secondary Outcome: Traditional Systemic Agent Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 12
Description: as for outcome 116
Time Frame: Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 88 | 20
doses | 2.0 (11.27) | 0.1 (0.31)

129. Secondary Outcome: Traditional Systemic Agent Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 18
Description: as for outcome 116
Time Frame: Month 18
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 63 | 19
doses | 0.6 (4.04) | 0.1 (0.23)

130. Secondary Outcome: Traditional Systemic Agent Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 24
Description: as for outcome 116
Time Frame: Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 63 | 16
doses | 1.4 (5.93) | 4.3 (15.02)

131. Secondary Outcome: Adalimumab Injection Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 3
Description: as for outcome 116
Time Frame: Month 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 9 | 224
doses | 0.0 (0.00) | 0.2 (0.54)

132. Secondary Outcome: Adalimumab Injection Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 6
Description: as for outcome 116
Time Frame: Month 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 17 | 207
doses | 1.2 (3.33) | 0.4 (1.37)

133. Secondary Outcome: Adalimumab Injection Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 12
Description: as for outcome 116
Time Frame: Month 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 28 | 177
doses | 0.9 (2.61) | 0.6 (1.59)

134. Secondary Outcome: Adalimumab Injection Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 18
Description: as for outcome 116
Time Frame: Month 18
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 32 | 160
doses | 0.1 (0.35) | 0.6 (2.36)

135. Secondary Outcome: Adalimumab Injection Patient Reported Treatment Compliance: Number of Missed Doses Since Last Visit Assessed at Month 24
Description: as for outcome 116
Time Frame: Month 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 29 | 154
doses | 0.0 (0.19) | 0.4 (1.17)

136. Secondary Outcome: Medical History: Number of Participants With Any Relevant Physical Changes Since the Last Visit at Month 3
Description: Changes in medical history were assessed by the treating physician since the last visit at Month 3, 6, 12, 18, and 24. A global assessment of physical changes per standard of care was recorded for each participant as "yes", "no", "not done" or missing.
Time Frame: Month 3
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 247 | 257
participants
  Yes | 76 | 88
  No | 167 | 162
  Not done | 4 | 6
  Missing | 0 | 1

137. Secondary Outcome: Medical History: Number of Participants With Any Relevant Physical Changes Since the Last Visit at Month 6
Description: as for outcome 136
Time Frame: Month 6
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 247
participants
  Yes | 75 | 75
  No | 145 | 168
  Not done | 2 | 3
  Missing | 1 | 1

138. Secondary Outcome: Medical History: Number of Participants With Any Relevant Physical Changes Since the Last Visit at Month 12
Description: as for outcome 136
Time Frame: Month 12
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 55 | 58
  No | 139 | 158
  Not done | 7 | 5
  Missing | 5 | 6

139. Secondary Outcome: Medical History: Number of Participants With Any Relevant Physical Changes Since the Last Visit at Month 18
Description: as for outcome 136
Time Frame: Month 18
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 171 | 199
participants
  Yes | 53 | 37
  No | 113 | 158
  Not done | 2 | 1
  Missing | 3 | 3

140. Secondary Outcome: Medical History: Number of Participants With Any Relevant Physical Changes Since the Last Visit at Month 24
Description: as for outcome 136
Time Frame: Month 24
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 51 | 41
  No | 111 | 143
  Not done | 2 | 8
  Missing | 4 | 2

141. Secondary Outcome: Concomitant Medication: Number of Participants With Any Changes in Psoriasis Medication/Treatment Since the Last Visit at Month 3
Description: Change in concomitant medication use by the participant was defined as any treatment, whether prescription or over the counter, used by the participant for psoriasis before and during the study. Details were recorded in the Case Report Form by the investigator and included dose, frequency, and duration of treatment and route. Change was assessed by treating physician per standard of care at Month 3, 6, 12, 18, and 24. A global assessment of change was recorded for each participant as "yes", "no", "not done" or missing.
Time Frame: Month 3
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 247 | 257
participants
  Yes | 106 | 88
  No | 139 | 166
  Not done | 1 | 1
  Missing | 1 | 2

142. Secondary Outcome: Concomitant Medication: Number of Participants With Any Changes in Psoriasis Medication/Treatment Since the Last Visit at Month 6
Description: as for outcome 141
Time Frame: Month 6
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 223 | 257
participants
  Yes | 108 | 68
  No | 113 | 177
  Not done | 1 | 1
  Missing | 1 | 1

143. Secondary Outcome: Concomitant Medication: Number of Participants With Any Changes in Psoriasis Medication/Treatment Since the Last Visit at Month 12
Description: as for outcome 141
Time Frame: Month 12
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 206 | 227
participants
  Yes | 88 | 63
  No | 108 | 157
  Not done | 5 | 1
  Missing | 5 | 6

144. Secondary Outcome: Concomitant Medication: Number of Participants With Any Changes in Psoriasis Medication/Treatment Since the Last Visit at Month 18
Description: as for outcome 141
Time Frame: Month 18
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 171 | 199
participants
  Yes | 65 | 53
  No | 102 | 143
  Not done | 1 | 0
  Missing | 3 | 3

145. Secondary Outcome: Concomitant Medication: Number of Participants With Any Changes in Psoriasis Medication/Treatment Since the Last Visit at Month 24
Description: as for outcome 141
Time Frame: Month 24
Population: ITT population of participants who were available for assessment at this visit.
Measure: Number; unit: participants
Arm/Group | Topical/Traditional Systemic Agent | Adalimumab
Number analyzed (Participants) | 168 | 194
participants
  Yes | 71 | 44
  No | 93 | 145
  Not done | 0 | 3
  Missing | 4 | 2

ADVERSE EVENTS:
Time Frame: Safety was assessed with the incidence of treatment-emergent adverse events (AEs) as recorded by the treating physician through the spontaneously reported events during the 24 months of treatment. Serious adverse events were reported to AbbVie from the time the physician obtained the participant's authorization to use and disclose information (or the participant's informed consent) until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment.
Description: Safety analysis set included all participants enrolled in the study and who received at least 1 dose of study drug (N = 658).
Groups:
- Topical/Traditional: Participants who initiated treatment with a new topical agent that was not used before or already being treated with topical agent and not responding, thereby requiring a change of treatment type, frequency, or dose and all participants who initiated treatment with a new systemic agent that was not used before alone or in combination with topical agents.
Arm/Group | Topical/Traditional | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/330 | 1/328
Serious Adverse Events (participants affected / at risk) | 2/330 | 23/328
Other Adverse Events (participants affected / at risk) | 1/330 | 14/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical/Traditional (N=330) | Adalimumab (N=328)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (2)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1)
ABDOMINAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 2 (3)
FATIGUE (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 2 (3)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (2)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PAROTID ABSCESS (Infections and infestations) | 0 (0) | 1 (2)
PAROTITIS (Infections and infestations) | 0 (0) | 1 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BRAIN NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (2)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 (0) | 1 (1)
BREAST MASS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ARTHRODESIS (Surgical and medical procedures) | 0 (0) | 1 (1)
CARPAL TUNNEL DECOMPRESSION (Surgical and medical procedures) | 0 (0) | 1 (1)
HEART VALVE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (2)
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
NAIL OPERATION (Surgical and medical procedures) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical/Traditional (N=330) | Adalimumab (N=328)
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 0 (0) | 1 (1)
DRUG INEFFECTIVE (General disorders) | 1 (1) | 8 (10)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (2)
PAIN (General disorders) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 1 (2)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
NAIL BED INFLAMMATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2013-08-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT01387815/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT01387815/SAP_001.pdf